CLINICAL TRIAL: NCT06120101
Title: Examining the Effect of Foot Reflexology Massage on Seizure Frequency, Fatigue, Stress and Sleep Quality in Epilepsy Patients: Randomized Control Experimental Research
Brief Title: Reflexology on Seizure Frequency, Fatigue, Stress and Sleep Quality in Epilepsy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, NİHAN TÜRKOĞLU, Assist Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NihanTurkoglu
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Reflexology; Epilepsy; Fatigue; Stress
MeSH Terms: conditions — Epilepsy; Fatigue | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Reflexology will be applied in a total of 3 sessions and the final test will be applied to the patients by phone 24 hours after the last reflexology application. At the end of the study, 3 reflexology sessions and 2 test measurements will be performed on the experimental group. Each reflexology session takes approximately 30-40 minutes. Sessions will be performed in a private room within the neurology clinic, on ergonomic and repositionable beds. Each session started with the right foot and will continue with the left foot. Primary relaxation techniques will be applied to both feet, followed by reflexology techniques to all system organs.
  Interventions: Behavioral: Reflexology Massage
- Control (No Intervention): No application will be applied to the control group.

INTERVENTIONS:
Behavioral: Reflexology Massage — The researcher washed his hands with an antibacterial soap before cleaning the patient's feet. The feet were cleaned according to the patient's preference; To wash feet with water or use disposable wet cloth. The patients were placed in a supine position on the bed in the room and their joint points were supported. The researcher stood at the end of the patient's bed during treatment. Unscented sesame oil at room temperature was used to provide lubrication during reflexology. The application started with the patient's right foot. The foot was first relaxed by applying effleurage, shaking, rotation and stretching methods. During the application, the researcher used the fingers of the other hand while supporting the patient's foot with one hand, and the thumb and caterpillar technique was mostly used. In other applications, the index finger and other fingers were used. The training ended by applying solar plexus pressure to both feet.
  Arms: Experimental

SUMMARY:
Epilepsy is among the diseases that cause loss of neurological abilities regardless of any trauma. Reflexology is one of the complementary therapies based on activating the body's self-healing power through special hand techniques applied to the feet. It is known that there are positive changes in seizure frequency, fatigue, stress and sleep quality in epilepsy patients after reflexology. This study will be conducted to determine the effect of reflexology on seizure frequency, fatigue, stress and sleep quality in epilepsy patients.

DETAILED DESCRIPTION:
Individual interviews were conducted with epilepsy patients who applied to the neurology clinic of a university hospital where the research was conducted, and patients who met the inclusion criteria and agreed to participate in the study will be randomly included in the experiment.

Patients arriving on the first day of the week will be placed in the experimental group. In the following days, groups will be formed as one day experiment and one day control (Monday-experiment, Tuesday-control, Wednesday-experiment, Thursday-control, Friday-experiment). Data collection tools will be applied to the experimental and control group patients at the beginning and end of the study. Only reflexology massage will be applied to the experimental group, and no application will be applied to the control group. Data will be collected simultaneously with the control and experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Knowing the diagnosis of the disease
* Having not received reflexology therapy before
* Being literate in Turkish
* Conscious Open,
* Able to communicate verbally,
* Being 18 years or older

Exclusion Criteria:

* Pain starts while doing massage,
* Having an infection,
* High fever,
* Having clot problems in the leg veins,
* Having an acute (newly developing) disease (heart attack, fainting, etc.),
* Wounds in the application area,
* Patients in the first 3 months of pregnancy.
* Paraplegia or thrombosis
* Leg varicose veins or foot disease (open wound or fracture on the foot)
* Diagnosis of psychiatric disorder or dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Chalder Fatigue Scale (CFA) | two week
  Individuals' fatigue level was evaluated with the CSI developed by Trudie Chalder in 1993. CWS is an 11-item scale that evaluates the fatigue felt by individuals during the last month through self-report. CEX consists of physical fatigue and mental fatigue subscales. A four-point Likert scale is used in the evaluation.
Perceived Stress Scale (PSS) | Two week
  It was developed by Cohen, Kamarck & Mermelste in 1983, and its Cronbach Alpha value was found to be 0.86 in the reliability study. In this study, the scale adapted to Turkish by Bilge, Öğce, Genç and Oran (2007) was used, and the Cronbach Alpha value was found to be 0.81 in the reliability study. Three items of the scale prepared in a 5-point Likert type (0 never, 4 very often) are reverse-worded (items 4, 5, 6), and five items are literal (items 1, 2, 3, 7, 8). ). A total score of 0-32 is taken from the scale. It has two subscales: perceived stress (items 1, 2, 3, 7, 8) and perceived coping (items 4, 5, and 6). The scale is evaluated on both total score and subscale scores. A high total score means a high perceived stress level. High scores from the subscales are a negative situation.
Pittsburg Sleep Quality scale (PSQI) | Two week
  The scale developed by Buysse et al., Turkish reliability and validity study by Ağargün et al. (Ağargün MY, Kara H, 1996). Made by. The scale, which examines the individual's sleep quality in the last month, consists of 24 items. Each question is evaluated with a number from 0 to 3. The highest score that can be obtained from the scale is 21. An increase in the score obtained from the scale indicates that sleep quality is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Türkoğlu, Principal Investigator — Ataturk University
Locations (1):
- Nihan Türkoğlu, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No